CLINICAL TRIAL: NCT04242264
Title: A Double-Blind Placebo Controlled Randomized Phase 2 Trial to Evaluate the Safety, Reactogenicity and Immunogenicity of a Live-Attenuated Shigella Sonnei Vaccine, WRSs2 and Determine Its Efficacy in a Challenge Model of S. Sonnei 53G in Healthy Adults
Brief Title: Phase 2 Shigella Vaccine and Challenge
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 17-0112
Record Dates: First submitted 2020-01-23; First posted 2020-01-27 (Actual); Results first posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2023-12-07

CONDITIONS: Immunisation; Shigella Infection
Keywords: Challenge; Double-blind; Efficacy; Healthy Adults; Immunogenicity; Live-attenuated Shigella sonnei Vaccine; Phase 2 Trial; Placebo-controlled; Protective efficacy; Randomized; Reactogenicity; Safety; Shigella sonnei 53G Challenge; WRSs2
MeSH Terms: conditions — Dysentery, Bacillary

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1 (Experimental): Vaccine: 1 ml of saline containing10^6 or 5X10^5 cfu of the WRSs2 vaccine in 30 ml of sterile normal saline administered orally on Day 1 and Day 29. Challenge: 1 ml of S. sonnei 53G challenge in 30 ml of sterile saline administered orally on Day 57. N=40
  Interventions: Biological: Shigella sonnei strain 53G; Biological: WRSs2
- Arm 2 (Experimental): Placebo + Vaccine: 30 ml of sterile normal saline placebo administered orally on Day 1 and 1 ml of saline containing 10^6 cfu of the WRSs2 vaccine in 30 ml of sterile normal saline administered orally on Day 29. Challenge: 1 ml of S. sonnei 53G challenge in 30ml of sterile saline administered orally on Day 57. N=40
  Interventions: Other: Placebo; Biological: Shigella sonnei strain 53G; Biological: WRSs2
- Arm 3 (Placebo Comparator): Placebo: 31 ml of sterile normal saline placebo administered orally on Day 1 and Day 29. Challenge: 1 ml of S. sonnei 53G challenge in 30 ml of sterile saline administered orally on Day 57. N=40
  Interventions: Other: Placebo; Biological: Shigella sonnei strain 53G

INTERVENTIONS:
Other: Placebo — 0.9% Sterile Normal Saline, USP
  Arms: Arm 2; Arm 3
Biological: Shigella sonnei strain 53G — 1.5 x 10^3 Colony Forming Units (cfu) Shigella sonnei 53G, a virulent strain of wildtype Shigella sonnei
Biological: WRSs2 — 10^6 Colony Forming Units (cfu) dose of an oral live-attenuated Shigella sonnei vaccine candidate derived from a virulent S. sonnei strain Moseley (WRSs2)-a live, attenuated vaccine that has been manufactured under cGMP conditions at the WRAIR PBF
  Arms: Arm 1; Arm 2

SUMMARY:
This is a trial to evaluate the safety, reactogenicity, immunogenicity and efficacy of a 10^6 cfu dose of an oral live-attenuated S. sonnei vaccine candidate, WRSs2, in up to 120 healthy males and non-pregnant females aged 18-49, inclusive. This is a two-phase study, an outpatient WRSs2 vaccination phase and an inpatient S. sonnei 53G challenge phase. After the initiation of the study, two participants had Grade 3 diarrhea and/or vomiting in the days following vaccination. The vaccination dose was reduced to 5X10^5, enrollment was changed to 2 arms and randomized 2:1 (vaccine: placebo). Participants with morbid obesity were excluded and weight loss medications prohibited. The Primary Objective of this study is to estimate combined vaccine efficacy of 2 doses of WRSs2 (10^6 cfu or 5X10^5 cfu) in preventing shigellosis, following challenge with S. sonnei strain 53G.

DETAILED DESCRIPTION:
This is a double-blind, placebo controlled, randomized study to test the safety, reactogenicity, immunogenicity and efficacy of up to a 10^6 cfu dose of an oral live-attenuated S. sonnei vaccine (WRSs2) to protect against shigellosis after a targeted oral challenge with S. sonnei 53G, a virulent strain of S. sonnei. Up to 120 subjects, healthy males and non-pregnant females aged 18-49, will be enrolled and randomized in this study. Using the 10^6 CFU dose, subjects were randomized 1:1:1 into one of three vaccination arms to receive 2 doses of study agent 28 days apart. Arm 1 received 2 doses of WRSs2, Arm 2 received placebo followed by WRSs2 and Arm 3 received 2 doses of placebo. Twenty-eight (+2) days after the second dose of study agent, subjects were admitted to the inpatient unit and given an oral challenge of approximately 1500 cfu of 53G. The goal was to have 90 subjects (30 per arm) receive a challenge dose of 53G. The study duration is approximately 24 months with subject participation duration approximately 8 months.

After the initiation of the study, two participants had Grade 3 diarrhea and/or vomiting in the days following vaccination. The vaccination dose was reduced to 5X10^5, enrollment was changed to 2 arms and randomized 2:1 (vaccine: placebo). Participants with morbid obesity were excluded and weight loss medications prohibited.

The Primary Objective of this study is to estimate combined vaccine efficacy of 2 doses of WRSs2 (10^6 cfu or 5X10^5 cfu) in preventing shigellosis, following challenge with S. sonnei strain 53G. The Secondary Objectives are to:1) Estimate vaccine efficacy of 1 dose of 10^6 cfu, 2 doses of 10^6 cfu, and 2 doses of 5x10^5 cfu of WRSs2 in preventing shigellosis following challenge with S. sonnei strain 53G. 2) Evaluate the safety of WRSs2; 3) Evaluate immune responses following vaccination (immunogenicity) with WRSs2 and after challenge with S. sonnei strain 53G by serum anti-LPS and anti-Invaplex IgG and IgA by ELISA; 4) Determine fecal shedding of S. sonnei after WRSs2 vaccination and 53G challenge by qualitative stool culture.

ELIGIBILITY:
Inclusion Criteria:

1. Provide informed consent prior to initiation of any study procedures.
2. Are able to understand and comply with planned study procedures and be available for all study visits.
3. Is 18-49 years of age inclusive and in sufficiently good health* to be safely enrolled in this study as determined by medical history, medication use, and abbreviated physical exam.

   *Good health is defined by the absence of any exclusionary medical conditions. If the subject has another current, ongoing medical condition, the condition cannot meet any of the following criteria: 1) first diagnosed within 3 months of enrollment; 2) is worsening in terms of clinical outcome in last 6 months; or 3) involves need for medication that may pose a risk to subject's safety or impede assessment of adverse events or immunogenicity if they participate in the study. Topical, nasal, and inhaled medications (with the exception of inhaled corticosteroids as outlined in the Subject Exclusion Criteria, herbals, vitamins, and supplements are permitted.
4. Oral temperature is less than 100.4 degrees Fahrenheit.
5. Pulse is 50 to 100 beats per minute (bpm), inclusive.
6. Systolic blood pressure is 90 to 140 mmHg, inclusive.
7. Diastolic blood pressure is 55 to 90 mmHg, inclusive.
8. Females of childbearing potential** may enroll if subject has practiced adequate contraception*** = / > 30 days prior to enrollment and agrees to continue adequate contraception for the entire study.

   **Child-bearing potential is defined as not sterilized via tubal ligation, bilateral oophorectomy, salpingectomy, hysterectomy, or successful Essure(R) placement (permanent, non-surgical, non-hormonal sterilization) with documented radiological confirmation test at least 90 days after the procedure, and still menstruating or <1 year of the last menses if menopausal.

   ***Adequate contraception includes; non-male sexual relationships, abstinence from sexual intercourse with a male partner, monogamous relationship with vasectomized partner who has been vasectomized for 180 days or more prior to the subject enrollment, barrier methods such as condoms or diaphragms with spermicide, effective intrauterine devices, NuvaRing(R), and licensed hormonal methods such as implants, injectables, or oral contraceptives ("the pill").
9. Females of childbearing potential must have a negative urine or serum pregnancy test within 24 hours prior to enrollment.
10. Drug screen for opiates is negative.
11. BMI (Body Mass Index) between 18 and 40kg/m^2.

Exclusion Criteria:

1. Have any disease or medical condition that, in the opinion of the site principal investigator or appropriate sub-investigator, is a contraindication to study participation****.

   **** Including acute or chronic disease or medical condition that would place the subject at an unacceptable risk of injury, render the subject unable to meet the requirements of the protocol, or may interfere with the evaluation of responses or the subject's successful completion of this trial. These include:
   1. History of inflammatory bowel disease (IBD) (including ulcerative colitis, Crohn's disease, indeterminate colitis, or celiac disease).
   2. Irritable bowel syndrome (IBS) within the past 12 months or any active uncontrolled gastrointestinal disorders or diseases as assessed by the investigator. Including: symptoms or evidence of active gastritis or gastroesophageal reflux disease, gastric surgery or gastric acid hyper-secretory disorders (e.g., Zollinger-Ellison syndrome), gastrointestinal obstruction, ileus, gastric retention, bowel perforation, toxic colitis, persistent infectious gastroenteritis, persistent or chronic diarrhea of unknown etiology, Clostridium difficile infection.
   3. Known active neoplastic disease (Non-melanoma, treated, skin cancers are permitted), a history of any hematologic malignancy, or have used anticancer chemotherapy/radiation therapy (cytotoxic) within 3 years prior to study enrollment.
   4. Personal or family history of reactive arthritis.
   5. Reported history of HIV, Hepatitis B, or Hepatitis C
   6. History of immunodeficiency due to congenital or hereditary causes, underlying illness or treatment.
2. Positive serology results for HLA-B27, HIV, HBsAg, or HCV antibodies.
3. Have clinically significant abnormalities as determined by study investigator in other screening laboratory tests, as outlined in the protocol.
4. Have participated in a previous Shigella challenge study or reports having received vaccination for Shigella previously.
5. Have a previously laboratory confirmed case of disease caused by S. sonnei or serology positive (>1:2500) for anti S. sonnei LPS IgG ELISA titer at screening.
6. Has a history of diarrhea in the 14 days prior to enrollment.
7. Have fewer than 3 stools per week or more than 3 stools per day as the usual frequency.
8. Recent history/current use of immunosuppressive/immunomodulating disease therapy.
9. Known hypersensitivity to ciprofloxacin or trimethoprim-sulfamethoxazole; sodium bicarbonate; or any components of vaccine, placebo, or challenge material.
10. Received or plan to receive a licensed live vaccine within 30 days prior to enrollment.
11. Received or plan to receive a licensed, inactivated, Coronavirus disease 2019 (COVID-19) vaccine or an influenza vaccine within +-7 days from receipt of study product.
12. Have a history of severe reactions following previous immunization with any licensed or unlicensed vaccine.
13. Received Ig or other blood products (with exception of Rho D Ig) within 90 days prior to enrollment.
14. Have taken oral or parenteral (including intra-articular) corticosteroids of any dose, or high-dose inhaled corticosteroids**within 30 days prior to enrollment.

    ** High-dose defined per age as using inhaled high dose per reference chart Estimated Comparative Daily Dosages https://www.nhlbi.nih.gov/files/docs/guidelines/asthma_qrg.pdf
15. Have taken systemic antibiotics within 7 days prior to enrollment.
16. Have taken prescription and/or OTC medication containing loperamide, acetaminophen, aspirin, ibuprofen, or other non-steroidal anti-inflammatory < / = 48 hours prior to enrollment.
17. Have a history of alcohol or drug abuse within 1 year prior to enrollment.
18. Have been hospitalized for psychiatric illness, history of suicide attempt, or confinement for danger to self or others within 5 years prior to enrollment.
19. Work or plan to work in either a health care setting, day care center, or as a food handler or have known daily contact with individuals with possible increased susceptibility****** to Shigella within 14 days after discharge from inpatient challenge.

    ****** Immunocompromised, elderly persons aged 70 years or more, diapered individuals, persons with disabilities, children < 2 years old, a woman known to be pregnant or nursing, or anyone with diminished immunity. Known daily contact includes contact at home, school, day-care, nursing home, or similar places.
20. Are pregnant, breastfeeding or plan to become pregnant or breastfeed at any given time during the study.
21. Have fever or an acute illness******* as determined by the site principal investigator or appropriate sub-investigator, within 72 hours prior to enrollment.

    ******* An acute illness which is nearly resolved with only minor residual symptoms remaining is allowable if, in the opinion of the site principal investigator or appropriate sub-investigator, the residual symptoms will not interfere with the ability to assess safety parameters as required by the protocol
22. Received an experimental agent (including vaccine, drug, biologic, device, blood product, or medication, other than from participation in this trial) within 30 days prior to the first study vaccination or expect to receive an investigational product during the study period which might affect safety or assessment of study endpoints.
23. Taking prescription or over-the-counter medication for weight reduction.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2022-10-12 (Actual); Primary Completion 2024-03-11 (Actual); Study Completion 2024-07-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - The Hope Clinic of Emory University, Decatur, Georgia
  - Cincinnati Children's Hospital Medical Center Vaccine Research Center, Cincinnati, Ohio

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were healthy males and non-pregnant females, 18-49 years inclusive at the time of first vaccination, who met all eligibility criteria. They were recruited from the general population at the participating study sites. Participants were enrolled between 11Oct2022 and 09Jan2024.
Groups:
- WRSs2 + WRSs2 (10^6 Cfu): 10^6 colony forming units (cfu) of WRSs2 administered orally as a 31 mL suspension on Day 1 and Day 29, followed by challenge with 1.5x10^3 cfu of wild type Shigella sonnei (S. sonnei) 53G administered orally as a 31 mL suspension on Day 57.
  WRSs2 is a live-attenuated S. sonnei vaccine candidate derived from the wild type S. sonnei "Moseley" strain. The lyophilized WRSs2 vaccine was manufactured under current good manufacturing practice (cGMP) at the Walter Reed Army Institute of Research (WRAIR) Pilot Bioproduction Facility (PBF). Lyophilized WRSs2 vaccine was reconstituted and suspended in 0.9% sterile normal saline prior to administration.
  Challenge strain 53G is a virulent S. sonnei strain initially isolated from a child with diarrhea in Tokyo. The lyophilized 53G was manufactured under cGMP at WRAIR PBF. Lyophilized 53G was reconstituted and suspended in 0.9% sterile normal saline prior to administration.
- WRSs2 + WRSs2 (5x10^5 Cfu): 5x10^5 colony forming units (cfu) of WRSs2 administered orally as a 31 mL suspension on Day 1 and Day 29, followed by challenge with 1.5x10^3 cfu of wild type Shigella sonnei (S. sonnei) 53G administered orally as a 31 mL suspension on Day 57.
  WRSs2 is a live-attenuated S. sonnei vaccine candidate derived from the wild type S. sonnei "Moseley" strain. The lyophilized WRSs2 vaccine was manufactured under current good manufacturing practice (cGMP) at the Walter Reed Army Institute of Research (WRAIR) Pilot Bioproduction Facility (PBF). Lyophilized WRSs2 vaccine was reconstituted and suspended in 0.9% sterile normal saline prior to administration.
  Challenge strain 53G is a virulent S. sonnei strain initially isolated from a child with diarrhea in Tokyo. The lyophilized 53G was manufactured under cGMP at WRAIR PBF. Lyophilized 53G was reconstituted and suspended in 0.9% sterile normal saline prior to administration.
- Placebo + WRSs2 (10^6 Cfu): Placebo administered orally as a 31 mL solution on Day 1, 10^6 colony forming units (cfu) of WRSs2 administered orally as a 31 mL suspension on Day 29, and challenge with 1.5x10^3 cfu of wild type Shigella sonnei (S. sonnei) 53G administered orally as a 31 mL suspension on Day 57.
  WRSs2 is a live-attenuated S. sonnei vaccine candidate derived from the wild type S. sonnei "Moseley" strain. The lyophilized WRSs2 vaccine was manufactured under current good manufacturing practice (cGMP) at the Walter Reed Army Institute of Research (WRAIR) Pilot Bioproduction Facility (PBF). Lyophilized WRSs2 vaccine was reconstituted and suspended in 0.9% sterile normal saline prior to administration.
  Placebo is 0.9% sterile normal saline of United States Pharmacopeia (USP) grade.
  Challenge strain 53G is a virulent S. sonnei strain initially isolated from a child with diarrhea in Tokyo. The lyophilized 53G was manufactured under cGMP at WRAIR PBF. Lyophilized 53G was reconstituted and suspended in 0.9% sterile normal saline prior to administration.
- Placebo + Placebo: Placebo administered orally as a 31 mL solution on Day 1 and Day 29, followed by challenge with 1.5x10^3 cfu of wild type Shigella sonnei (S. sonnei) 53G administered orally as a 31 mL suspension on Day 57.
  Placebo is 0.9% sterile normal saline of United States Pharmacopeia (USP) grade.
  Challenge strain 53G is a virulent S. sonnei strain initially isolated from a child with diarrhea in Tokyo. The lyophilized 53G was manufactured under cGMP at WRAIR PBF. Lyophilized 53G was reconstituted and suspended in 0.9% sterile normal saline prior to administration.
Period: Overall Study
Arm/Group | WRSs2 + WRSs2 (10^6 Cfu) | WRSs2 + WRSs2 (5x10^5 Cfu) | Placebo + WRSs2 (10^6 Cfu) | Placebo + Placebo
Started | 22 | 26 | 23 | 37
Completed | 19 | 24 | 22 | 36
Not Completed | 3 | 2 | 1 | 1
Not completed — Lost to Follow-up | 2 | 2 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population includes all enrolled participants.
Groups:
- WRSs2 + WRSs2 (10^6 Cfu): 10^6 colony forming units (cfu) of WRSs2 administered orally as a 31 mL suspension on Day 1 and Day 29, followed by challenge with 1.5x10^3 cfu of wild type Shigella sonnei (S. sonnei) 53G administered orally as a 31 mL suspension on Day 57.
- WRSs2 + WRSs2 (5x10^5 Cfu): 5x10^5 colony forming units (cfu) of WRSs2 administered orally as a 31 mL suspension on Day 1 and Day 29, followed by challenge with 1.5x10^3 cfu of wild type Shigella sonnei (S. sonnei) 53G administered orally as a 31 mL suspension on Day 57.
- Placebo + WRSs2 (10^6 Cfu): Placebo administered orally as a 31 mL solution on Day 1, 10^6 colony forming units (cfu) of WRSs2 administered orally as a 31 mL suspension on Day 29, and challenge with 1.5x10^3 cfu of wild type Shigella sonnei (S. sonnei) 53G administered orally as a 31 mL suspension on Day 57.
- Placebo + Placebo: Placebo administered orally as a 31 mL solution on Day 1 and Day 29, followed by challenge with 1.5x10^3 cfu of wild type Shigella sonnei (S. sonnei) 53G administered orally as a 31 mL suspension on Day 57.
- Total: Total of all reporting groups
Arm/Group | WRSs2 + WRSs2 (10^6 Cfu) | WRSs2 + WRSs2 (5x10^5 Cfu) | Placebo + WRSs2 (10^6 Cfu) | Placebo + Placebo | Total
Number analyzed (Participants) | 22 | 26 | 23 | 37 | 108
Age, Continuous [Mean (Standard Deviation); unit: years] | 32 (7.7) | 31.8 (7.5) | 38.3 (8.3) | 31.2 (7.8) | 33 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 11 | 12 | 22 | 58
  Male | 9 | 15 | 11 | 15 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 1 | 4 | 9
  Not Hispanic or Latino | 20 | 24 | 22 | 33 | 99
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 6 | 9 | 14 | 33
  White | 17 | 18 | 12 | 18 | 65
  More than one race | 0 | 1 | 2 | 4 | 7
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 22 | 26 | 23 | 37 | 108
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 32.69 (8.33) | 28.29 (5.17) | 29.17 (5.93) | 29.72 (6.89) | 29.86 (6.74)

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Participants With Shigellosis Following Challenge With Shigella Sonnei 53G Through Day 63 in the Pooled Group of Participants Receiving Two Doses of 10^6 Cfu or 5x10^5 Cfu of WRSs2 Compared to Participants Receiving Two Doses of Placebo.
Description: Following study vaccination on Days 1 and 29, participants were admitted to an inpatient facility and challenged with Shigella sonnei strain 53G on Day 57. From challenge through Day 63, all stools passed by challenged participants were graded for consistency, all grade 3-5* stools were visually assessed for gross blood, and all gross blood-containing stools were confirmed via hemoccult test. A blinded endpoint review committee of independent Shigella experts determined whether shigellosis occurred for each participant based on number, weight, consistency, and hemoccult-positive status of stools, along with the presence of additional enteric symptoms.
  *Stool consistency was graded according to the following scale: 1 = Normal stool (best outcome); 2 = Soft stool; 3 = Loose stool; 4 = Watery stool; 5 = Rice water (worst outcome).
Time Frame: Day 57 through Day 63
Population: The Full Analysis Population includes all randomized participants who were challenged with complete data for the primary efficacy endpoint. Participants will be analyzed according to the study arm to which they were randomized.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Groups:
- WRSs2 + WRSs2 (10^6 Cfu or 5x10^5 Cfu): 10^6 colony forming units (cfu) or 5x10^5 cfu of WRSs2 administered orally as a 31 mL suspension on Day 1 and Day 29, followed by challenge with 1.5x10^3 cfu of wild type Shigella sonnei (S. sonnei) 53G administered orally as a 31 mL suspension on Day 57.
Arm/Group | WRSs2 + WRSs2 (10^6 Cfu or 5x10^5 Cfu) | Placebo + Placebo
Number analyzed (Participants) | 34 | 26
proportion of participants | 0.09 [0.03 to 0.23] | 0.81 [0.62 to 0.91]
Statistical Analysis 1: Comparison: WRSs2 + WRSs2 (10^6 Cfu or 5x10^5 Cfu) vs Placebo + Placebo; The null hypothesis is that the absolute vaccine efficacy (VE) of preventing shigellosis is zero. The alternative hypothesis is that the absolute VE is greater than zero; Test type: Superiority — A two-sided Chi-squared test with alpha=0.05 was used to test the null hypothesis that the vaccine efficacy is zero, which is equivalent to testing that the relative risk of shigellosis is one; p < 0.001, Chi-squared; Vaccine efficacy = 0.89, 95% CI 2-sided [0.71 to 0.96] — Vaccine efficacy was calculated as 1 - relative risk of shigellosis, where relative risk = probability of shigellosis in WRSs2 group / probability of shigellosis in placebo group. A Wilson (Score) CI was calculated for the vaccine efficacy estimate

2. Secondary Outcome: The Proportion of Participants With Shigellosis Following Challenge With S. Sonnei 53G Through Day 63 in Participants Receiving 1 Dose of 10^6 Cfu, 2 Doses of 10^6 Cfu, or 2 Doses of 5x10^5 Cfu of WRSs2 Compared to Those Receiving Two Doses of Placebo.
Description: as for outcome 1
Time Frame: Day 57 through Day 65
Population: The Full Analysis Population includes all randomized participants who were challenged with complete data for the primary efficacy endpoint. Participants were analyzed according to the study arm to which they were randomized.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | WRSs2 + WRSs2 (10^6 Cfu) | WRSs2 + WRSs2 (5x10^5 Cfu) | Placebo + WRSs2 (10^6 Cfu) | Placebo + Placebo
Number analyzed (Participants) | 16 | 18 | 13 | 26
proportion of participants | 0.19 [0.07 to 0.43] | 0 [0 to 0.18] | 0 [0 to 0.23] | 0.81 [0.62 to 0.91]
Statistical Analysis 1: Comparison: WRSs2 + WRSs2 (10^6 Cfu) vs Placebo + Placebo; Test type: Other — Vaccine efficacy was calculated as 1 - relative risk of shigellosis, where relative risk = probability of shigellosis in WRSs2 group / probability of shigellosis in placebo group. A Wilson (Score) CI was calculated for the vaccine efficacy estimate, but no formal hypothesis test was performed; Vaccine efficacy = 0.77, 95% CI 2-sided [0.44 to 0.92]
Statistical Analysis 2: Comparison: WRSs2 + WRSs2 (5x10^5 Cfu) vs Placebo + Placebo; Test type: Other — [test comment as in outcome 2, analysis 1]; Vaccine efficacy = 1.00, 95% CI 2-sided [0.78 to 1.00]
Statistical Analysis 3: Comparison: Placebo + WRSs2 (10^6 Cfu) vs Placebo + Placebo; Test type: Other — [test comment as in outcome 2, analysis 1]; Vaccine efficacy = 1.00, 95% CI 2-sided [0.71 to 1.00]

3. Secondary Outcome: Number and Percentage of Participants With Solicited Systemic Adverse Events (AEs) Through 7 Days After Each Study Vaccination.
Description: Systemic solicited adverse events (AEs) were collected pre-vaccination, 90 minutes post-vaccination, and then daily for 7 days after each vaccination using a memory aid and graded on a scale of 0 (none), 1 (mild), 2 (moderate) and 3 (severe). Systemic events include fever, headache, arthralgia, nausea, pain/abdominal cramps, fatigue/malaise, myalgia, anorexia/loss of appetite, chills, vomiting, and diarrhea.
Time Frame: Day 1 through Day 8, Day 29 through Day 36
Population: The Safety Population includes all participants who received at least one dose of study vaccination. The number of participants analyzed for solicited systemic AEs after each vaccination reflects the number of participants in the Safety Population who received the corresponding vaccination. Participants were analyzed according to the study product actually received, not necessarily the study product to which a participant was randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | WRSs2 + WRSs2 (10^6 Cfu) | WRSs2 + WRSs2 (5x10^5 Cfu) | Placebo + WRSs2 (10^6 Cfu) | Placebo + Placebo
Number analyzed (Participants) | 22 | 26 | 22 | 38
Participants
  Post first vaccination (Day 1 through Day 8) | 17 | 22 | 11 | 27
  Post second vaccination (Day 29 through Day 36): number analyzed (Participants) | 18 | 23 | 16 | 30
  Post second vaccination (Day 29 through Day 36) | 13 | 17 | 11 | 22

4. Secondary Outcome: Number and Percentage of Participants With Vaccine-related Unsolicited AEs Through 28 Days Post Last Vaccination
Description: ICH E6 defines an AE as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product regardless of its causal relationship to the study treatment. FDA defines an AE as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related.
  An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of medicinal (investigational) product. The occurrence of an AE may come to the attention of study personnel during study visits and interviews of a study recipient presenting for medical care, or upon review by a study monitor.
  An AE is considered related if there is a reasonable possibility that the study product caused the AE. Reasonable possibility means that there is evidence to suggest a causal relationship between the study product and the AE.
Time Frame: Day 1 through Day 57
Population: The Safety Population includes all participants who received at least one dose of study vaccination. Participants were analyzed according to the study product actually received, not necessarily the study product to which a participant was randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | WRSs2 + WRSs2 (10^6 Cfu) | WRSs2 + WRSs2 (5x10^5 Cfu) | Placebo + WRSs2 (10^6 Cfu) | Placebo + Placebo
Number analyzed (Participants) | 22 | 26 | 22 | 38
Participants | 2 | 5 | 2 | 0

5. Secondary Outcome: Number and Percentage of Participants With SAEs Through Study Day 180 or Until Resolution or Stabilization Even if This Extends Beyond the Study-reporting Period.
Description: An AE or suspected adverse reaction is considered "serious" if, in the view of either the investigator or sponsor, it results in any of the following outcomes:
  * Death
  * A life-threatening AE
  * Inpatient hospitalization or prolongation of existing hospitalization
  * A persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions
  * A congenital anomaly/birth defect
  * Important medical events that may not result in death, be life-threatening, or require hospitalizations may be considered serious when, based upon appropriate medical judgment they may jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the outcomes listed in this definition.
Time Frame: Day 1 through Day 180
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | WRSs2 + WRSs2 (10^6 Cfu) | WRSs2 + WRSs2 (5x10^5 Cfu) | Placebo + WRSs2 (10^6 Cfu) | Placebo + Placebo
Number analyzed (Participants) | 22 | 26 | 22 | 38
Participants | 0 | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With >=4-fold Rise From Pre-vaccination in Anti-LPS (Lipopolysaccharide) IgG (Immunoglobulin G)
Description: Serum was collected pre-challenge at Day 1 (pre-dose 1), Day 15 (post-dose 1), Day 29 (pre-dose 2), Day 43 (post-dose 2), and Day 56 (post-dose 2) to assess IgG antibody response against LPS (a Shigella sonnei antigen) as measured by Enzyme Linked ImmunoSorbent Assay (ELISA). The number of participants with at least a 4-fold rise in antibody titer on each post-vaccination day as compared to pre-dose 1 is reported.
Time Frame: Day 15, Day 29, Day 43, and Day 56
Population: The Immunogenicity Population consists of all participants who received any study product and for whom immunogenicity endpoint data are available. Participants were analyzed according to the study product actually received, not necessarily the study product to which a participant was randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | WRSs2 + WRSs2 (10^6 Cfu) | WRSs2 + WRSs2 (5x10^5 Cfu) | Placebo + WRSs2 (10^6 Cfu) | Placebo + Placebo
Number analyzed (Participants) | 22 | 25 | 22 | 36
Participants
  Day 15 (Post-Dose 1) | 16 | 19 | 0 | 0
  Day 29 (Pre-Dose 2): number analyzed (Participants) | 22 | 24 | 20 | 34
  Day 29 (Pre-Dose 2) | 13 | 12 | 0 | 0
  Day 43 (Post-Dose 2): number analyzed (Participants) | 21 | 24 | 18 | 35
  Day 43 (Post-Dose 2) | 9 | 9 | 9 | 0
  Day 56 (Post-Dose 2): number analyzed (Participants) | 20 | 23 | 18 | 33
  Day 56 (Post-Dose 2) | 8 | 7 | 7 | 0

7. Secondary Outcome: Number of Participants With >=4-fold Rise From Pre-vaccination in Anti-Invaplex IgG (Immunoglobulin G)
Description: Serum was collected pre-challenge at Day 1 (pre-dose 1), Day 15 (post-dose 1), Day 29 (pre-dose 2), Day 43 (post-dose 2), and Day 56 (post-dose 2) to assess IgG antibody response against Invaplex (a Shigella sonnei antigen complex) as measured by Enzyme Linked ImmunoSorbent Assay (ELISA). The number of participants with at least a 4-fold rise in antibody titer on each post-vaccination day as compared to pre-dose 1 is reported.
Time Frame: Day 15, Day 29, Day 43, and Day 56
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | WRSs2 + WRSs2 (10^6 Cfu) | WRSs2 + WRSs2 (5x10^5 Cfu) | Placebo + WRSs2 (10^6 Cfu) | Placebo + Placebo
Number analyzed (Participants) | 22 | 25 | 22 | 36
Participants
  Day 15 (Post-Dose 1) | 16 | 13 | 0 | 0
  Day 29 (Pre-Dose 2): number analyzed (Participants) | 22 | 24 | 20 | 34
  Day 29 (Pre-Dose 2) | 16 | 11 | 0 | 0
  Day 43 (Post-Dose 2): number analyzed (Participants) | 21 | 24 | 18 | 35
  Day 43 (Post-Dose 2) | 14 | 10 | 9 | 1
  Day 56 (Post-Dose 2): number analyzed (Participants) | 20 | 23 | 18 | 33
  Day 56 (Post-Dose 2) | 11 | 9 | 9 | 1

8. Secondary Outcome: Number of Participants With >=4-fold Rise From Pre-vaccination in Anti-LPS (Lipopolysaccharide) IgA (Immunoglobulin A)
Description: Serum was collected pre-challenge at Day 1 (pre-dose 1), Day 15 (post-dose 1), Day 29 (pre-dose 2), Day 43 (post-dose 2), and Day 56 (post-dose 2) to assess IgA antibody response against LPS (a Shigella sonnei antigen) as measured by Enzyme Linked ImmunoSorbent Assay (ELISA). The number of participants with at least a 4-fold rise in antibody titer on each post-vaccination day as compared to pre-dose 1 is reported.
Time Frame: Day 15, Day 29, Day 43, and Day 56
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | WRSs2 + WRSs2 (10^6 Cfu) | WRSs2 + WRSs2 (5x10^5 Cfu) | Placebo + WRSs2 (10^6 Cfu) | Placebo + Placebo
Number analyzed (Participants) | 22 | 25 | 22 | 36
Participants
  Day 15 (Post-Dose 1) | 19 | 24 | 0 | 0
  Day 29 (Pre-Dose 2): number analyzed (Participants) | 22 | 24 | 20 | 34
  Day 29 (Pre-Dose 2) | 12 | 18 | 0 | 1
  Day 43 (Post-Dose 2): number analyzed (Participants) | 21 | 24 | 18 | 35
  Day 43 (Post-Dose 2) | 9 | 12 | 13 | 1
  Day 56 (Post-Dose 2): number analyzed (Participants) | 20 | 23 | 18 | 33
  Day 56 (Post-Dose 2) | 6 | 6 | 10 | 0

9. Secondary Outcome: Number of Participants With >=4-fold Rise From Pre-vaccination in Anti-Invaplex IgA (Immunoglobulin A)
Description: Serum was collected pre-challenge at Day 1 (pre-dose 1), Day 15 (post-dose 1), Day 29 (pre-dose 2), Day 43 (post-dose 2), and Day 56 (post-dose 2) to assess IgA antibody response against Invaplex (a Shigella sonnei antigen complex) as measured by Enzyme Linked ImmunoSorbent Assay (ELISA). The number of participants with at least a 4-fold rise in antibody titer on each post-vaccination day as compared to pre-dose 1 is reported.
Time Frame: Day 15, Day 29, Day 43, and Day 56
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | WRSs2 + WRSs2 (10^6 Cfu) | WRSs2 + WRSs2 (5x10^5 Cfu) | Placebo + WRSs2 (10^6 Cfu) | Placebo + Placebo
Number analyzed (Participants) | 22 | 25 | 22 | 36
Participants
  Day 15 (Post-Dose 1) | 20 | 24 | 0 | 0
  Day 29 (Pre-Dose 2): number analyzed (Participants) | 22 | 24 | 20 | 34
  Day 29 (Pre-Dose 2) | 14 | 21 | 0 | 1
  Day 43 (Post-Dose 2): number analyzed (Participants) | 21 | 24 | 18 | 35
  Day 43 (Post-Dose 2) | 16 | 15 | 13 | 3
  Day 56 (Post-Dose 2): number analyzed (Participants) | 20 | 23 | 18 | 33
  Day 56 (Post-Dose 2) | 9 | 9 | 13 | 2

10. Secondary Outcome: Maximum Anti-LPS (Lipopolysaccharide) and Anti-Invaplex Serum IgG (Immunoglobulin G) and IgA (Immunoglobulin A) Titer Post-vaccination Through Day 56
Description: Serum was collected post-vaccination and pre-challenge at Day 15 (post-dose 1), Day 29 (pre-dose 2), Day 43 (post-dose 2), and Day 56 (post-dose 2) to assess IgG and IgA antibody responses against LPS and Invaplex (Shigella sonnei antigens) as measured by Enzyme Linked ImmunoSorbent Assay (ELISA). The maximum titer per participant between first vaccination (Day 1) and challenge (Day 57) is summarized by study arm via geometric mean and 95% confidence interval.
Time Frame: Day 15 through Day 56
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | WRSs2 + WRSs2 (10^6 Cfu) | WRSs2 + WRSs2 (5x10^5 Cfu) | Placebo + WRSs2 (10^6 Cfu) | Placebo + Placebo
Number analyzed (Participants) | 22 | 25 | 22 | 36
titer
  Anti-LPS IgG | 1758.6 [1081.3 to 2860.1] | 1837.9 [1206.2 to 2800.5] | 997.4 [624.4 to 1593.2] | 423.8 [323.2 to 555.7]
  Anti-Invaplex IgG | 5467.2 [3373.0 to 8861.6] | 5571.5 [3924.5 to 7909.7] | 1873.0 [1078.0 to 3254.4] | 1371.6 [970.3 to 1938.8]
  Anti-LPS IgA | 1062.3 [593.6 to 1901.1] | 1026.7 [710.4 to 1483.9] | 341.7 [186.3 to 626.9] | 110.1 [85.6 to 141.6]
  Anti-Invaplex IgA | 1814.9 [956.3 to 3444.3] | 1472.3 [1005.5 to 2155.9] | 426.0 [221.0 to 821.3] | 110.1 [80.5 to 150.6]

11. Secondary Outcome: Peak Fold-rise From Pre-vaccination in Anti-LPS (Lipopolysaccharide) and Anti-Invaplex Serum IgG (Immunoglobulin G) and IgA (Immunoglobulin A) Titer
Description: Serum was collected post-vaccination and pre-challenge at Day 15 (post-dose 1), Day 29 (pre-dose 2), Day 43 (post-dose 2), and Day 56 (post-dose 2) to assess IgG and IgA antibody responses against LPS and Invaplex (Shigella sonnei antigens) as measured by Enzyme Linked ImmunoSorbent Assay (ELISA). The peak fold-rise is calculated per participant at the maximum titer value post-vaccination (and before challenge) compared to pre-vaccination and is summarized by study arm via geometric mean fold-rise and 95% confidence interval.
Time Frame: Day 15 through Day 56
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise from pre-vaccination
Arm/Group | WRSs2 + WRSs2 (10^6 Cfu) | WRSs2 + WRSs2 (5x10^5 Cfu) | Placebo + WRSs2 (10^6 Cfu) | Placebo + Placebo
Number analyzed (Participants) | 22 | 25 | 22 | 36
fold rise from pre-vaccination
  Anti-LPS IgG | 5.0 [3.4 to 7.4] | 4.1 [3.1 to 5.5] | 3.2 [1.8 to 5.7] | 1.2 [1.1 to 1.3]
  Anti-Invaplex IgG | 7.8 [4.9 to 12.3] | 3.3 [2.3 to 4.7] | 3.1 [2.0 to 4.9] | 1.3 [1.1 to 1.4]
  Anti-LPS IgA | 12.0 [7.0 to 20.7] | 11.8 [8.4 to 16.6] | 4.3 [2.3 to 7.8] | 1.2 [1.0 to 1.4]
  Anti-Invaplex IgA | 20.6 [11.3 to 37.4] | 14.3 [9.5 to 21.6] | 6.2 [3.2 to 12.0] | 1.4 [1.1 to 1.7]

12. Secondary Outcome: Number of Participants With >=4-fold Rise From Pre-challenge in Anti-LPS (Lipopolysaccharide) IgG (Immunoglobulin G)
Description: Serum was collected post-challenge at Days 64, 71, 85, and 113 to assess IgG antibody response against LPS (a Shigella sonnei antigen) as measured by Enzyme Linked ImmunoSorbent Assay (ELISA). The number of participants with at least a 4-fold rise in antibody titer on each post-challenge day as compared to pre-challenge is reported.
Time Frame: Day 64, Day 71, Day 85, and Day 113
Population: This analysis includes participants in the Immunogenicity Population who were challenged. The Immunogenicity Population consists of all participants who received any study product and for whom immunogenicity endpoint data are available. Participants were analyzed according to the study product actually received, not necessarily the study product to which a participant was randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | WRSs2 + WRSs2 (10^6 Cfu) | WRSs2 + WRSs2 (5x10^5 Cfu) | Placebo + WRSs2 (10^6 Cfu) | Placebo + Placebo
Number analyzed (Participants) | 16 | 18 | 13 | 26
Participants
  Day 64 | 1 | 0 | 0 | 3
  Day 71: number analyzed (Participants) | 15 | 18 | 12 | 26
  Day 71 | 2 | 1 | 0 | 20
  Day 85: number analyzed (Participants) | 16 | 18 | 12 | 26
  Day 85 | 1 | 1 | 0 | 16
  Day 113: number analyzed (Participants) | 14 | 18 | 12 | 26
  Day 113 | 1 | 0 | 1 | 12

13. Secondary Outcome: Number of Participants With >=4-fold Rise From Pre-challenge in Anti-Invaplex IgG (Immunoglobulin G)
Description: Serum was collected post-challenge at Days 64, 71, 85, and 113 to assess IgG antibody response against Invaplex (a Shigella sonnei antigen complex) as measured by Enzyme Linked ImmunoSorbent Assay (ELISA). The number of participants with at least a 4-fold rise in antibody titer on each post-challenge day as compared to pre-challenge is reported.
Time Frame: Day 64, Day 71, Day 85, and Day 113
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | WRSs2 + WRSs2 (10^6 Cfu) | WRSs2 + WRSs2 (5x10^5 Cfu) | Placebo + WRSs2 (10^6 Cfu) | Placebo + Placebo
Number analyzed (Participants) | 16 | 18 | 13 | 26
Participants
  Day 64 | 1 | 0 | 0 | 4
  Day 71: number analyzed (Participants) | 15 | 18 | 12 | 26
  Day 71 | 4 | 1 | 0 | 20
  Day 85: number analyzed (Participants) | 16 | 18 | 12 | 26
  Day 85 | 1 | 0 | 0 | 15
  Day 113: number analyzed (Participants) | 14 | 18 | 12 | 26
  Day 113 | 0 | 0 | 0 | 14

14. Secondary Outcome: Number of Participants With >=4-fold Rise From Pre-challenge in Anti-LPS (Lipopolysaccharide) IgA (Immunoglobulin A)
Description: Serum was collected post-challenge at Days 64, 71, 85, and 113 to assess IgA antibody response against LPS (a Shigella sonnei antigen) as measured by Enzyme Linked ImmunoSorbent Assay (ELISA). The number of participants with at least a 4-fold rise in antibody titer on each post-challenge day as compared to pre-challenge is reported.
Time Frame: Day 64, Day 71, Day 85, and Day 113
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | WRSs2 + WRSs2 (10^6 Cfu) | WRSs2 + WRSs2 (5x10^5 Cfu) | Placebo + WRSs2 (10^6 Cfu) | Placebo + Placebo
Number analyzed (Participants) | 16 | 18 | 13 | 26
Participants
  Day 64 | 2 | 0 | 1 | 13
  Day 71: number analyzed (Participants) | 15 | 18 | 12 | 26
  Day 71 | 7 | 7 | 1 | 24
  Day 85: number analyzed (Participants) | 16 | 18 | 12 | 26
  Day 85 | 1 | 2 | 0 | 17
  Day 113: number analyzed (Participants) | 14 | 18 | 12 | 26
  Day 113 | 0 | 0 | 0 | 7

15. Secondary Outcome: Number of Participants With >=4-fold Rise From Pre-challenge in Anti-Invaplex IgA (Immunoglobulin A)
Description: Serum was collected post-challenge at Days 64, 71, 85, and 113 to assess IgA antibody response against Invaplex (a Shigella sonnei antigen complex) as measured by Enzyme Linked ImmunoSorbent Assay (ELISA). The number of participants with at least a 4-fold rise in antibody titer on each post-challenge day as compared to pre-challenge is reported.
Time Frame: Day 64, Day 71, Day 85, and Day 113
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | WRSs2 + WRSs2 (10^6 Cfu) | WRSs2 + WRSs2 (5x10^5 Cfu) | Placebo + WRSs2 (10^6 Cfu) | Placebo + Placebo
Number analyzed (Participants) | 16 | 18 | 13 | 26
Participants
  Day 64 | 3 | 0 | 0 | 13
  Day 71: number analyzed (Participants) | 15 | 18 | 12 | 26
  Day 71 | 5 | 8 | 1 | 22
  Day 85: number analyzed (Participants) | 16 | 18 | 12 | 26
  Day 85 | 3 | 3 | 0 | 22
  Day 113: number analyzed (Participants) | 14 | 18 | 12 | 26
  Day 113 | 0 | 0 | 0 | 9

16. Secondary Outcome: Maximum Anti-LPS (Lipopolysaccharide) and Anti-Invaplex Serum IgG (Immunoglobulin G) and IgA (Immunoglobulin A) Titer Post-challenge Through Day 113
Description: Serum was collected post-challenge at Days 64, 71, 85, and 113 to assess IgG and IgA antibody responses against LPS and Invaplex (Shigella sonnei antigens) as measured by Enzyme Linked ImmunoSorbent Assay (ELISA). The maximum titer per participant between challenge (Day 57) and Day 113 is summarized by study arm via geometric mean and 95% confidence interval.
Time Frame: Day 64 through Day 113
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | WRSs2 + WRSs2 (10^6 Cfu) | WRSs2 + WRSs2 (5x10^5 Cfu) | Placebo + WRSs2 (10^6 Cfu) | Placebo + Placebo
Number analyzed (Participants) | 16 | 18 | 13 | 26
titer
  Anti-LPS IgG | 1233.8 [709.0 to 2147.1] | 1175.8 [805.7 to 1715.9] | 843.8 [528.9 to 1346.2] | 2145.3 [1419.7 to 3241.5]
  Anti-Invaplex IgG | 4525.5 [2245.5 to 9120.5] | 4887.8 [3237.6 to 7379.2] | 1600.0 [717.4 to 3568.2] | 6400.0 [4273.9 to 9583.8]
  Anti-LPS IgA | 436.2 [211.3 to 900.4] | 400.0 [229.7 to 696.5] | 275.4 [166.7 to 454.9] | 1044.4 [697.0 to 1564.9]
  Anti-Invaplex IgA | 590.7 [219.3 to 1591.0] | 565.7 [301.8 to 1060.4] | 323.2 [225.9 to 462.3] | 1557.9 [929.8 to 2610.3]

17. Secondary Outcome: Peak Fold-rise From Pre-challenge in Anti-LPS (Lipopolysaccharide) and Anti-Invaplex Serum IgG (Immunoglobulin G) and IgA (Immunoglobulin A) Titer
Description: Serum was collected post-challenge at Days 64, 71, 85, and 113 to assess IgG and IgA antibody responses against LPS and Invaplex (Shigella sonnei antigens) as measured by Enzyme Linked ImmunoSorbent Assay (ELISA). The peak fold-rise is calculated per participant at the maximum titer value post-challenge compared to pre-challenge and is summarized by study arm via geometric mean fold-rise and 95% confidence interval.
Time Frame: Day 64 through Day 113
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise from pre-challenge
Arm/Group | WRSs2 + WRSs2 (10^6 Cfu) | WRSs2 + WRSs2 (5x10^5 Cfu) | Placebo + WRSs2 (10^6 Cfu) | Placebo + Placebo
Number analyzed (Participants) | 16 | 18 | 13 | 26
fold rise from pre-challenge
  Anti-LPS IgG | 1.8 [1.3 to 2.6] | 1.2 [0.9 to 1.5] | 1.1 [0.8 to 1.6] | 6.1 [4.0 to 9.4]
  Anti-Invaplex IgG | 1.9 [1.3 to 2.8] | 1.2 [0.9 to 1.5] | 1.0 [0.7 to 1.3] | 5.8 [3.7 to 9.0]
  Anti-LPS IgA | 2.6 [1.5 to 4.4] | 2.2 [1.3 to 3.6] | 1.2 [0.7 to 2.0] | 12.9 [8.2 to 20.3]
  Anti-Invaplex IgA | 2.5 [1.4 to 4.5] | 2.5 [1.4 to 4.5] | 0.8 [0.5 to 1.3] | 18.3 [10.6 to 31.5]

18. Secondary Outcome: Number of Participants Shedding Vaccine Strain in Their Stool by Culture Prior to Challenge
Description: Stool samples collected at baseline and on Days 4, 8, 15, 29, 32, 36, 43, and 56 were cultured for shedding of Shigella sonnei. For this outcome measure, "baseline" is considered the last day at which culture results were available pre-vaccination (may be at screening visit or Day 1). In the event a subject was unable to produce a bulk stool, rectal swabs were collected for culture.
Time Frame: Baseline (day of last culture prior to dose 1) through Day 56
Population: The Shedding Analysis Population consists of all participants who received any study product. Participants were analyzed according to the study product they actually received, not necessarily the study product to which a participant was randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | WRSs2 + WRSs2 (10^6 Cfu) | WRSs2 + WRSs2 (5x10^5 Cfu) | Placebo + WRSs2 (10^6 Cfu) | Placebo + Placebo
Number analyzed (Participants) | 22 | 26 | 22 | 38
Participants
  Baseline (Pre-Dose 1) | 0 | 0 | 0 | 0
  Day 4 (Post-Dose 1) | 15 | 14 | 0 | 0
  Day 8 (Post-Dose 1): number analyzed (Participants) | 22 | 25 | 22 | 38
  Day 8 (Post-Dose 1) | 15 | 19 | 0 | 0
  Day 15 (Post-Dose 1): number analyzed (Participants) | 21 | 25 | 21 | 36
  Day 15 (Post-Dose 1) | 3 | 10 | 0 | 0
  Day 29 (Pre-Dose 2): number analyzed (Participants) | 22 | 24 | 20 | 35
  Day 29 (Pre-Dose 2) | 4 | 6 | 0 | 0
  Day 32 (Post-Dose 2): number analyzed (Participants) | 16 | 23 | 16 | 30
  Day 32 (Post-Dose 2) | 7 | 5 | 9 | 0
  Day 36 (Post-Dose 2): number analyzed (Participants) | 17 | 23 | 16 | 30
  Day 36 (Post-Dose 2) | 3 | 4 | 9 | 0
  Day 43 (Post-Dose 2): number analyzed (Participants) | 17 | 23 | 16 | 30
  Day 43 (Post-Dose 2) | 2 | 1 | 6 | 1
  Day 56 (Post-Dose 2): number analyzed (Participants) | 16 | 23 | 16 | 29
  Day 56 (Post-Dose 2) | 0 | 2 | 4 | 0

19. Secondary Outcome: Number of Participants Shedding 53G in Their Stool by Culture Post-challenge
Description: Stool samples collected on Day 57 (post-challenge) through Day 65 were cultured for shedding of Shigella sonnei strain 53G. In the event a subject was unable to produce a bulk stool, rectal swabs were collected for culture.
Time Frame: Day 57 (post-challenge) through Day 65
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | WRSs2 + WRSs2 (10^6 Cfu) | WRSs2 + WRSs2 (5x10^5 Cfu) | Placebo + WRSs2 (10^6 Cfu) | Placebo + Placebo
Number analyzed (Participants) | 16 | 18 | 13 | 26
Participants
  Day 57 | 0 | 0 | 3 | 0
  Day 58 | 0 | 1 | 2 | 5
  Day 59 | 4 | 3 | 2 | 19
  Day 60 | 6 | 3 | 4 | 19
  Day 61 | 9 | 6 | 5 | 13
  Day 62 | 7 | 4 | 3 | 13
  Day 63 | 0 | 1 | 1 | 0
  Day 64 | 0 | 0 | 0 | 0
  Day 65 | 0 | 0 | 0 | 0

20. Secondary Outcome: Mean Duration of Shedding Vaccine Strain Post-vaccination Through Day 56 by Culture.
Description: Stool samples collected on Day 1 (post-vaccination) and on Days 4, 8, 15, 29, 32, 36, 43, and 56 were cultured for shedding of Shigella sonnei. In the event a subject was unable to produce a bulk stool, rectal swabs were collected for culture.
  The duration of shedding is evaluated from the day of the initial positive culture result to the day of the last positive qualitative or quantitative culture, regardless of intermittent negative results.
Time Frame: Day 1 (post-vaccination) through Day 56
Population: This analysis includes participants in the Shedding Analysis Population with detected Shigella shedding post vaccination and prior to challenge. The Shedding Analysis Population consists of all participants who received any study product. Participants were analyzed according to the study product they actually received, not necessarily the study product to which a participant was randomized.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | WRSs2 + WRSs2 (10^6 Cfu) | WRSs2 + WRSs2 (5x10^5 Cfu) | Placebo + WRSs2 (10^6 Cfu) | Placebo + Placebo
Number analyzed (Participants) | 14 | 22 | 11 | 1
days | 21.9 (14.6) | 15.9 (15.0) | 13.3 (10.3) | 1.0 (NA) — Only one participant experienced shedding, so standard deviation of shedding duration could not be calculated.

21. Secondary Outcome: Mean Duration of Shedding 53G Post-challenge Through Day 65 by Culture.
Description: Stool samples collected on Day 57 (post-challenge) through Day 65 were cultured for shedding of Shigella sonnei strain 53G. In the event a subject was unable to produce a bulk stool, rectal swabs were collected for culture.
  The duration of shedding is evaluated from the day of the initial positive culture result to the day of the last positive qualitative or quantitative culture, regardless of intermittent negative results.
Time Frame: Day 57 (post-challenge) through Day 65
Population: This analysis includes participants in the Full Analysis Population with detected Shigella shedding post challenge. The Full Analysis Population includes all randomized participants who were challenged with complete data for the primary efficacy endpoint. Participants were analyzed according to the study arm to which they were randomized.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | WRSs2 + WRSs2 (10^6 Cfu) | WRSs2 + WRSs2 (5x10^5 Cfu) | Placebo + WRSs2 (10^6 Cfu) | Placebo + Placebo
Number analyzed (Participants) | 10 | 8 | 8 | 23
days | 2.6 (1.3) | 2.6 (1.2) | 2.5 (1.3) | 3.1 (1.3)

ADVERSE EVENTS:
Time Frame: Solicited adverse events (AEs) and clinical safety laboratory AEs were collected after each study vaccination through Day 8 after vaccination. Unsolicited non-serious AEs were reported from first study vaccination through approximately Day 57. Serious adverse events (SAEs) were collected from first study vaccination through approximately Day 180 or until resolution or stabilization of the SAE.
Description: Adverse events are presented by actual study product received. One participant randomized to the "Placebo + WRSs2 (10^6 cfu)" Arm was actually administered Placebo + Placebo. For adverse event results, this participant is counted among those at risk in the "Placebo + Placebo" Arm.
Arm/Group | WRSs2 + WRSs2 (10^6 Cfu) | WRSs2 + WRSs2 (5x10^5 Cfu) | Placebo + WRSs2 (10^6 Cfu) | Placebo + Placebo
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/26 | 0/22 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/26 | 0/22 | 0/38
Other Adverse Events (participants affected / at risk) | 21/22 | 25/26 | 19/22 | 36/38
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | WRSs2 + WRSs2 (10^6 Cfu) (N=22) | WRSs2 + WRSs2 (5x10^5 Cfu) (N=26) | Placebo + WRSs2 (10^6 Cfu) (N=22) | Placebo + Placebo (N=38)
Tachycardia (Cardiac disorders) | 1 (2) | 0 (0) | 3 (4) | 15 (20)
Abdominal pain (Gastrointestinal disorders) | 6 (8) | 12 (18) | 7 (9) | 12 (13)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1) | 1 (1)
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 6 (6)
Nausea (Gastrointestinal disorders) | 5 (5) | 7 (9) | 6 (7) | 13 (17)
Chills (General disorders) | 5 (6) | 10 (12) | 5 (6) | 5 (5)
Malaise (General disorders) | 12 (19) | 16 (22) | 9 (12) | 18 (25)
Pyrexia (General disorders) | 1 (1) | 5 (8) | 1 (1) | 10 (10)
Viral infection (Infections and infestations) | 2 (2) | 2 (2) | 3 (3) | 2 (2)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Blood pressure diastolic decreased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 2 (2)
Blood pressure systolic increased (Investigations) | 3 (3) | 0 (0) | 1 (2) | 4 (5)
Decreased appetite (Metabolism and nutrition disorders) | 8 (8) | 11 (13) | 4 (4) | 10 (11)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (11) | 7 (8) | 4 (6) | 8 (9)
Myalgia (Musculoskeletal and connective tissue disorders) | 8 (10) | 8 (9) | 4 (6) | 8 (10)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 13 (19) | 18 (25) | 10 (15) | 23 (30)
Diastolic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (5)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (3):
  • Study Protocol (2023-09-14): https://cdn.clinicaltrials.gov/large-docs/64/NCT04242264/Prot_001.pdf
  • Statistical Analysis Plan (2024-11-12): https://cdn.clinicaltrials.gov/large-docs/64/NCT04242264/SAP_002.pdf
  • Informed Consent Form (2023-10-12): https://cdn.clinicaltrials.gov/large-docs/64/NCT04242264/ICF_000.pdf